CLINICAL TRIAL: NCT00488930
Title: Characteristics of Dendritic Cells Before and After Gastric Banding
Status: Terminated | Type: Observational
Why Stopped: Terminated due to a lack of recruitment and decision by the PI not to continue.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Santiago Horgan, Professor of Surgery, University of California, San Diego
Other Study IDs: 070685; Internal Funding; NIH MED 1736
Record Dates: First submitted 2007-06-11; First posted 2007-06-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Morbid Obesity; Hyperglycemia; Diabetes Mellitus
Keywords: Obesity; Hyperglycemia; Diabetes Mellitus Type I; Diabetes Mellitus Type II
MeSH Terms: conditions — Obesity, Morbid; Hyperglycemia; Diabetes Mellitus; Obesity; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational — data collection ONLY

SUMMARY:
A research study to find out more about a specific white blood cell called a dendritic cell. These cells are found in a layer of fat in the body called the omentum. The omentum is a layer of fat that covers the bowels (intestines) and protects them.

The purpose of this study is to allow us to compare dendritic cells in normal weight individuals to the dendritic cells of people who are extremely overweight. These cells will be collected from the omentum, the layer of fat that covers and protects the bowels (intestines), from the mesentery, which is another layer of fat that surrounds the intestines directly, and from the subcutaneous tissue, which is the layer of fat just under the skin.

DETAILED DESCRIPTION:
Obesity continues to be a major source of morbidity and mortality in the United States. The association between obesity and type II diabetes is well known. Several studies suggest that fat may generate a low grade inflammatory response that may be responsible for the metabolic changes in obese patients. More specifically, a certain type of white blood cell that causes inflammation called a dendritic cell has been found in high concentrations in omental fat. This cell has not been extensively studied in human patients with morbid obesity, though it may play a central role in the development of insulin resistance. Aside from weight loss, the surgical treatment of obesity also results in a decrease in the markers of inflammation. Many of the comorbidities of morbid obesity improve or are cured. Laparoscopic adjustable gastric banding is safer than other gastric bypass procedures and results in similar amounts of weight loss after 2 years postoperatively.

Much of the work regarding dendritic cells in human subjects has been in patients with Crohn's disease. Both the cytokine profile and characteristics of the dendritic cells have been extensively studied in Crohn's patients, but not in obese individuals. In addition to this, these cells have not been re-evaluated after a period of weight loss.

A more detailed analysis of the inflammation of obesity and its subsequent resolution with weight loss will contribute to the growing body of information on this subject. Further work will lend insight into the pathogenesis of the comorbidities of obesity and may contribute to uncovering potential treatments for these illnesses. Dendritic cells have been extensively studied in animal models. We now know specific cell surface markers and signaling pathways for these cells, their responses to stimulating factors, and their ability to secrete anti-inflammatory cytokines such as IL-10. We hope to translate these findings to humans.

It is now recognized that chronic low-grade inflammation is the critical element leading to insulin resistance in insulin target cells. The evidence for this is substantial, including consistent measurements of elevated inflammatory markers in plasma from insulin resistance/diabetic humans and rodents. This concept was further established by the recent discovery that obese adipose tissue contains large numbers of resident macrophages. In fact, in the lean state, about 10% of all the cell types within adipose tissue consist of macrophages, and this number can go as high as 50% in obesity. Furthermore, FACS sorting of adipose tissue macrophages based on surface markers, has indicated that it is a subpopulation of macrophages which accounts for this remarkable increase. This subpopulation involves macrophages which are positive for F4/80, CD11B and CD11C and are, therefore, dendritic-like in their phenotype. There are also reports in the literature which suggests that visceral adipose tissue may be particularly "inflamed" compared to subcutaneous adipose tissue and that increased macrophage infiltration and inflammatory markers are expressed in visceral fat. More recent evidence, in which the macrophage inflammatory pathway is specifically disabled, in knock-out mice, conclusively demonstrates that the macrophage can be the initiating or orchestrating cell type responsible for the inflammatory response which ultimately leads to systemic insulin resistance.

These concepts will be assessed in using the subcutaneous and visceral fat samples obtained under this protocol. The adipose tissue samples will be collagenase digested to release all of the adipocytes and non-adipocyte cell types within the tissue. Using differential centrifugation and filtration, the stromal vascular fraction (SVF) will be separated from the adipocytes. The SVF contains the macrophages, and these cells will undergo FACS analysis based on the expression of F4/80, CD11B and CD11C to determine the absolute number of macrophages within a given adipose tissue sample, and the proportion of classical macrophages versus dendritic cell-like macrophages. The cells will then be sorted, and inflammatory marker expression will be measured in the classical macrophages (F4/80 positive, CD11B positive, but CD11C negative) versus the dendritic-like cells (F480 positive, CD11B positive, and CD11C positive). This analysis will involve direct measurement of cytokine expression by these cells (TNF, IL-1, and IL-6) as well as PCR-based measurements of mRNA expression of inflammatory pathway components. These measurements will be performed on the subcutaneous and visceral adipose tissue obtained at the time of the initial surgery, as well as on the subcutaneous adipose tissue samples at follow up after weight reduction.

ELIGIBILITY:
Inclusion Criteria:

* For gastric banding subjects to qualify for study inclusion, subjects have to have a BMI ranging from 33-40. Currently a BMI of 33 is our lower level of acceptable for bypass. Subjects with a BMI>40 will be excluded because their fat cells are very large and therefore fragile and unsuitable for research use.

Control Group:

* All adult subjects 18 years or greater being seen in the minimally invasive surgery clinic for elective laparoscopic surgery will also be screened.
* These will be subjects who are non-obese (BMI<30) and undergoing laparoscopic surgery for a different indication such as hernia repair or cholecystectomy. These will be patients who are undergoing elective procedures to minimize the impact an acute inflamed abdomen may have on the fat cells.

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant will be excluded from this study. Gastric banding cannot not be performed on pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects being treated for obesity at this institution
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Measure changes in dendritic cells at baseline, 6 months and 1 year following weight loss | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Horgan, MD, Principal Investigator — UCSD; Jerrold M Olefsky, MD, Study Director — UCSD
Locations (1):
- UCSD Medical Center, San Diego, California, United States